CLINICAL TRIAL: NCT02188875
Title: Wearable Sensor/Device With Website (Fitbit One) and SMS Text Messaging Prompts to Increase Physical Activity in Overweight/Obese Adults: A Randomized Controlled Pilot Trial
Brief Title: Fitbit One and Text Messaging Prompts to Promote Physical Activity in Overweight/Obese Adults
Acronym: TXT2BFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Carol Vassiliadis Family (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 130024
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Health Behavior; Obesity
Keywords: Fitbit One; wearable sensor; wearable device; web-based intervention; SMS text messages; randomized controlled trial; physical activity; behavioral intervention; text message prompts; text messaging; technology; exercise
MeSH Terms: conditions — Health Behavior; Obesity; Motor Activity | interventions — Wearable Electronic Devices; Blood Glucose Self-Monitoring; Professional Autonomy; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Text Messages & Fitbit One (Experimental): All study participants were provided a Fitbit One to facilitate self-monitoring of PA. Those who were randomly assigned to the intervention group were asked to indicate 3 preferred times of the day to receive text message prompts to do PA throughout the 6-week study period.
  Interventions: Behavioral: SMS Text Messages & Fitbit One
- Fitbit One Only (Active Comparator): An active control group was also provided the Fitbit One to facilitate self-monitoring of PA throughout the 6-week study period.
  Interventions: Behavioral: Fitbit One Only

INTERVENTIONS:
Behavioral: SMS Text Messages & Fitbit One — The primary aim was to test text-messaging in its basic form to prompt physical activity. A secondary aim was to examine the effects of the Fitbit One.
  Other Names: Fitbit One; SMS text-messaging; SMS text-messages; wearable sensor; wearable device; text message reminders; text message prompts; Actigraph GT3X+; self-monitoring; self-regulation; physical activity; website; tracker; mobile application; mobile app; MVPA; fairly active minutes; very active minutes
  Arms: SMS Text Messages & Fitbit One
Behavioral: Fitbit One Only — Active controls received a Fitbit One to facilitate self-monitoring (and no text messages)
  Other Names: Fitbit One; wearable sensor; wearable device; text message reminders; text message prompts; Actigraph GT3X+; self-monitoring; self-regulation; physical activity; website; tracker; mobile application; mobile app; MVPA; fairly active minutes; very active minutes
  Arms: Fitbit One Only

SUMMARY:
Previous studies suggest self-regulatory techniques including self-monitoring, and SMS text-messaging as an intervention modality, can modify health behaviors including physical activity (PA). The primary purpose of this study was to examine change in objectively measured PA in a randomized controlled pilot trial that tested a wearable sensor/device (Fitbit One) for self-monitoring and SMS text-messaging prompts to promote PA in overweight/obese adults. In a 2-group design, 67 participants were provided the Fitbit One and half were randomized to receive 3 daily SMS-based PA prompts. A Fitbit One was provided to facilitate self-monitoring with a wearable tracker for instant feedback and website of daily PA summaries. Outcome measures were number of steps and minutes of PA by intensity-level using two accelerometers: Actigraph GT3X+ (primary) at baseline and 6-week follow-up and Fitbit One (secondary) at baseline and weeks 1-6. The main hypothesis was that text messaging plus the Fitbit One would show a greater increase in steps and minutes of PA compared to only the Fitbit One at 6-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-69 years of age
* overweight or obese (otherwise healthy)
* does not meet recommended levels of PA (>150 min/wk of MVPA)
* owns a personal mobile phone and able to use SMS text-messaging
* owns a personal computer, has access to Internet, able to operate the Fitbit One
* fluent in English

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
steps per day (Actigraph GT3X+) | up to 6 weeks
  Number of steps per day was measured using Actigraph GT3X+ at baseline and 6-week follow-up

SECONDARY OUTCOMES:
Minutes per week of physical activity by intensity level (Actigraph GT3X+) | up to 6 weeks
  Moderate-to-vigorous intensity physical activity (MVPA) (min/wk) and total PA (min/wk) were assessed using Actigraph GT3X+ at baseline week and 6-week follow-up

OTHER OUTCOMES:
Physical activity levels (Fitbit One) | up to 6 weeks
  Physical activity by intensity level (i.e., fairly and very active minutes and total active minutes) were assessed using the Fitbit One throughout the entire duration of the study
Steps per a day (Fitbit One) | up to 6 weeks
  Steps per day were assessed using the Fitbit One throughout the entire duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wang, PhD, MPH, Principal Investigator — University of California, San Francisco; John Pierce, PhD, Study Chair — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

REFERENCES:
- See also: published manuscript of primary study results — http://online.liebertpub.com/doi/abs/10.1089/tmj.2014.0176